CLINICAL TRIAL: NCT05938439
Title: Evaluation of the Performance of MAgnetic Gastrointestinal Universal Septotome for Treatment of Candy Cane Syndrome
Acronym: MAGUS-CCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Brussel Medical Device Center (BMDC) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N2023/021
Record Dates: First submitted 2023-06-22; First posted 2023-07-10 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-06

CONDITIONS: Blind Loop Syndrome Postoperative; Candy Cane Syndrome
Keywords: candy cane syndrome; therapeutic endoscopy; steptotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): The procedure consists in Medical Device (MAGUS) placement by endoscopy under general anesthesia with fluoroscopic control.
  Interventions: Device: MAGUS placement

INTERVENTIONS:
Device: MAGUS placement — An upper endoscopy will be performed with the use of fluoroscopy under general anaesthesia with orotracheal intubation. The delivery system will be placed over a guidewire, under fluoroscopy. The main steps are the following:
  * Placement through the endoscope of a soft guidewire through the upper GI tract;
  * Insertion of the MAGUS system on the guidewire;
  * Advancement of the MAGUS system until proximal magnet reach the top of the septum;
  * Release and placement of the proximal magnet at the bottom of the septum, pouch side;
  * Meeting of the distal and proximal magnet on both sides of the septum, by pulling on the delivery system;
  * Release of the distal magnet and activate the retractable wire;
  * Insure that wire is not blocked and unblocked it if applicable.
  Endoscopy and contrast injection will be performed before and after placement to ensure the correct positioning of the magnets.

SUMMARY:
Candy cane syndrome (CCS) is an adverse event (AE) from gastrectomy or gastric bypass and end-to-side anastomosis to a jejunal loop. It seems to be predominantly mechanical, the afferent blind loop enlarge and becomes preferential passage of food. This food accumulated in the blind loop increase luminal pressure, causing dilatation, early satiety, fullness, pain, reflux, regurgitation, postprandial vomiting, weight loss, and, ultimately, inability to eat, leading to cachexia.Up to now, main treatment is laparoscopic revision which is invasive. Adverse events related this surgical procedure occurred in 13,3% of cases and substantial improvement only in 73.9%.

A first clinical study with MAGUS including oesophageal diverticulum (n=2) and CCS (n=14) has been performed to assess safety and feasibility of this new device. MAGUS is an implantable device which is placed endoscopically and which, by using pressure necrosis, entailed the marsupialization of the blind loop in less than 30 days. Substantial improvement was observed in all patient and only 7,1% of patients experience an adverse event possibly related to the device. This study aim therefore to assess the safety and performance of the endoscopic treatment of CCS using a new medical device: MAGUS.

This will be a single-center, open-label prospective, safety and performance study on 51 patients with Candy Cane Syndrome (CCS). Patients will be followed for 12 months after the procedure, with an enrolment period of 3 years.

After the screening, the following data will be collected and examinations and tests performed : physical Exam, medical history including CCS cause and treatment(s) history, weight, Eckart and dysphagia score, Quality of Life questionnaire (SF 12 and GERD HRQL), Main symptom selection (Nausea, Vomiting/regurgitation or pain), nausea VAS, vomiting, regurgitation VAS, pain VAS, barium swallow X-ray or endoscopic assessment of Candy Cane. Follow-up visits will be performed at 14 days, 28 days, 3 months and 12 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with candy cane syndrome based on clinical and endoscopic and/or radiologic assessment
* Patient has at least one of this 3 symptoms associated to CCS: pain, nausea, vomiting, regurgitation
* Patient agrees and is able to comply with the study procedures and provide written informed consent to participate in the study

Exclusion Criteria:

* Refractory stenosis of the UGI proximal to the septum
* Septum height smaller than 2 cm or higher than 8 cm
* Coagulation disorders.

  • Previous implantation of a magnetic-sensitive medical device (including active electronic implant, metallic stent, …).
* Dysphagia related to motility disorder
* Planned MRI in the following month (30 days) of intervention
* Condition that could compromise patient safety
* Patient who went through an abdominal surgery less than 8 weeks before implantation of the magnets
* Patient pregnant, breastfeeding or incapacitated
* Patient currently enrolled in another clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety related to the number of adverse event | During procedure (operative day) ; at 14 days of follow-up ; at 28 days of follow-up ; at 3 months of follow-up
  All adverse events device or procedure related will be captured
Performance on symptoms evolution | At baseline ; at 14 days of follow-up ; at 28 days of follow-up ; at 3 months of follow-up ; at 12 months of follow-up
  Evolution of pain will be assessed on a visual analog scale from 0 (= no symptom) to 10 (= severe symptom)
Performance on symptoms evolution | At baseline ; at 14 days of follow-up ; at 28 days of follow-up ; at 3 months of follow-up ; at 12 months of follow-up
  Evolution of nausea will be assessed on a visual analog scale from 0 (= no symptom) to 10 (= severe symptom)
Performance on symptoms evolution | At baseline ; at 14 days of follow-up ; at 28 days of follow-up ; at 3 months of follow-up ; at 12 months of follow-up
  Evolution of regurgitations/vomiting will be assessed on a visual analog scale from 0 (= no symptom) to 10 (= severe symptom)

SECONDARY OUTCOMES:
Safety : adverse event at mid and long term | After 3 months of implantation
  All adverse events will be reported
Safety : unplanned interventions | Within the year following device placement
  Number of unplanned interventions
Efficacy : patient's satisfaction with the therapy | At 3 and 12 months of follow-up
  Scored by a visual analogue scale from 0 (= not satisfied at all) to 5 (=very satisfied)
Efficacy : change in quality of life | At 28 days, 3 months and 12 months of follow-up
  Short-Form-12 score. A higher score indicates a better quality of life
Efficacy : dysphagia evolution | At 14 and 28 days, and at 3 and 12 months of follow-up
  Eckart score from 0 to 12. A higher score indicates more severe pathology.
Efficacy : dysphagia evolution | At 14 and 28 days, and at 3 and 12 months of follow-up
  Dysphagia score from 1 to 5. A higher score indicates more severe pathology.
Efficacy : weight evolution | At 14 and 28 days, and at 3 and 12 months of follow-up
  Weight measurment in kg

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire de Bruxelles - Hôpital Erasme, Brussels, Belgium

REFERENCES:
- [Background] Rio-Tinto R, Huberland F, Van Ouytsel P, Delattre C, Dugardeyn S, Cauche N, Delchambre A, Deviere J, Blero D. Magnet and wire remodeling for the treatment of candy cane syndrome: first case series of a new approach (with video). Gastrointest Endosc. 2022 Jun;95(6):1247-1253. doi: 10.1016/j.gie.2021.12.027. Epub 2022 Jan 1. PMID 34979115